CLINICAL TRIAL: NCT00086957
Title: Phase I/II Trial of ZD1839 (Iressa®), Trastuzumab (Herceptin®), and Docetaxel (Taxotere®) in Patients With erbB-2 (HER-2) Overexpressing, Stage IV Breast Carcinoma
Brief Title: Gefitinib, Trastuzumab, and Docetaxel in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03049; P30CA033572 (NIH); CHNMC-03049; ZENECA-1839US/0274; ZENECA-IRUSIRES0012; CDR0000371908 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; male breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Trastuzumab; Docetaxel; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ZD1839, Trastuzumab and Docetaxel (Experimental)
  Interventions: Biological: trastuzumab; Drug: docetaxel; Drug: gefitinib

INTERVENTIONS:
Biological: trastuzumab — Cycle 1 loading dose of 8 mg/kg, followed by 6 mg/kg every 3 weeks for subsequent cycles.
Drug: docetaxel — 75 mg/m2 every three weeks, or 60 mg/m2 every three weeks depending on study findings
Drug: gefitinib — 250 mg daily or 250 mg daily on days 2 through 14 depending on study findings

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining gefitinib and trastuzumab with docetaxel may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the best dose of docetaxel when given together with gefitinib and trastuzumab in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and efficacy of gefitinib, trastuzumab (Herceptin®), and docetaxel, in terms of time to disease progression, in patients with HER2/neu-overexpressing metastatic adenocarcinoma of the breast.

Secondary

* Determine the objective tumor response rate in patients treated with this regimen.
* Correlate expression and/or degree of phosphorylation of epidermal growth factor receptor, HER2/neu, c-fos, Akt, ERK½, P13K, p53, p21, and p27 with outcome in patients treated with this regimen.

OUTLINE: This is a phase I, multicenter, dose-escalation study of docetaxel followed by a phase II study. Patients are stratified according to trastuzumab (Herceptin®)-naive vs trastuzumab-failure.

* Phase I: Patients receive oral gefitinib once daily on days 2-14. Patients also receive trastuzumab* IV over 30-90 minutes and docetaxel IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

NOTE: *Trastuzumab is given at a higher dose (loading dose) in course 1 and then at a lower dose in subsequent courses.

Cohorts of 3-6 patients receive docetaxel at dose level 1. If no dose-limiting toxicity (DLT) is observed in the first cohort of 3 patients, the dose of docetaxel remains the same. If 1 DLT is observed in the first cohort of 3 patients, 3 additional patients are added (for a total of 6 patients) to dose level 1. If no further DLTs are observed at dose level 1, the dose of docetaxel remains the same. If 2 of 3 or 2 of 6 patients experience DLT at dose level 1, the dose of docetaxel is considered above the maximum tolerated dose (MTD) and is subsequently reduced. If 2 of 3 or 2 of 6 patients experience DLT at the reduced dose of docetaxel, the study is stopped.

* Phase II: Patients receive docetaxel at the MTD and gefitinib and trastuzumab as in phase I.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 3-76 patients will be accrued for this study within 26 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Metastatic disease
* HER-2/neu overexpression (3+ by immunohistochemistry OR 2+ by fluorescence in situ hybridization)
* Measurable or evaluable disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* AST and ALT < 2.5 times upper limit of normal (ULN) (5.0 times ULN in the presence of liver metastases)
* Bilirubin < 1.5 times ULN
* No unstable or uncompensated hepatic disease

Renal

* Creatinine < 1.6 mg/dL
* No unstable or uncompensated renal disease

Cardiovascular

* LVEF > 45% by echocardiogram or MUGA
* No prior New York Heart Association class I-IV heart disease
* No prolonged PR interval or atrioventricular block on ECG
* No unstable or uncompensated cardiac disease

Pulmonary

* No unstable or uncompensated respiratory disease
* No clinically active interstitial lung disease

  * Patients who are asymptomatic and have chronic stable radiographic changes are allowed

Immunologic

* No autoimmune disorders
* No conditions of immunosuppression
* No severe hypersensitivity to taxane or gefitinib or any of its excipients

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other prior or concurrent malignancy within the past 5 years except basal cell carcinoma or carcinoma in situ of the cervix
* No other severe or uncontrolled systemic disease
* No other acute or chronic medical condition that would preclude study participation
* No other significant clinical disorder or laboratory finding that would preclude study participation
* No psychiatric illness that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior adjuvant trastuzumab (Herceptin®) allowed if > 6 months elapsed before disease recurrence
* No prior trastuzumab for metastatic breast cancer
* No prior monoclonal antibodies directed at the epidermal growth factor receptor (EGFR)

Chemotherapy

* Prior adjuvant chemotherapy (or as first-line therapy for metastatic breast cancer) allowed
* Prior adjuvant taxane allowed if completed > 6 months before diagnosis of metastatic breast cancer
* No prior docetaxel for metastatic breast cancer

Endocrine therapy

* Prior adjuvant hormonal therapy (or as first-line therapy for metastatic breast cancer) allowed
* No concurrent hormonal therapy

  * Concurrent steroids allowed provided dose is stable

Radiotherapy

* Not specified

Surgery

* Fully recovered from prior oncologic or other major surgery
* No concurrent surgery within 7 days of gefitinib administration

Other

* Recovered from prior anticancer therapy (alopecia allowed)
* More than 30 days since prior non-approved drug or investigational agent
* No other prior EGFR-directed therapy (i.e., tyrosine kinase inhibitors)
* No concurrent use of any of the following medications:

  * Phenytoin
  * Carbamazepine
  * Barbiturates
  * Rifampin
  * Hypericum perforatum (St. John's wort)
* No other concurrent anticancer therapy
* No concurrent cardioprotective drugs
* No concurrent oral retinoids
* Concurrent participation in the City of Hope indium-labeled trastuzumab imaging study allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2004-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Somlo, MD, Principal Investigator — City of Hope Medical Center
Locations (6):
- United States (6):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Hematology Oncology Consultants-Hemet, Hemet, California
  - Breastlink Medical Group, Incorporated at Long Beach Memorial Medical Center, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - City of Hope Medical Group, Pasadena, California

REFERENCES:
- [Result] Somlo G, Koczywas M, Luu T, et al.: A phase I-II study of trastuzumab, gefitinib, and docetaxel as first line chemotherapy in patients with HER-2 overexpressing stage IV breast carcinoma. [Abstract] Breast Cancer Research and Treatment 94 (Suppl 1): A-2035, 2005.

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I - Docetaxel 75 mg/m^2: Subjects receive gefitinib 250 mg orally daily, trastuzumab 6 mg/kg intravenously every 3 weeks (after an initial dose of 8 mg/kg with cycle 1), and docetaxel 75 mg/m^2 intravenously every 3 weeks.
- Phase I - Docetaxel 60 mg/m^2; Phase II - Docetaxel 60 mg/m^2: Subjects receive gefitinib 250 mg orally daily or 250 mg daily on days 2 through 14 depending on study findings, trastuzumab 6 mg/kg intravenously every 3 weeks (after an initial dose of 8 mg/kg with cycle 1), and docetaxel 60 mg/m^2 intravenously every 3 weeks.
Period: Overall Study
Arm/Group | Phase I - Docetaxel 75 mg/m^2 | Phase I - Docetaxel 60 mg/m^2 | Phase II - Docetaxel 60 mg/m^2
Started | 2 | 7 | 22
Completed | 2 | 7 | 22
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Levels 1 & 2 - Docetaxel 60 & 75 mg/m^2: trastuzumab: Cycle 1 loading dose of 8 mg/kg, followed by 6 mg/kg every 3 weeks for subsequent cycles.
  docetaxel: 75 mg/m^2 every three weeks, or 60 mg/m^2 every three weeks depending on study findings
  gefitinib: 250 mg daily or 250 mg daily on days 2 through 14 depending on study findings
Arm/Group | Dose Levels 1 & 2 - Docetaxel 60 & 75 mg/m^2
Number analyzed (Participants) | 31
Age, Continuous [Mean (Full Range); unit: years] | 52 [34 to 67]
Gender [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Dose Limiting Toxicity in Phase I
Description: Dose Limiting Toxicity (DLT) defined as any treatment-related grade 3 or greater except for hematological toxicities which must be grade 4. Interstitial Lung Disease (ILD) related to treatment should be considered as a DLT regardless of the grade.
Time Frame: 4 weeks from start of treatment, up to 2 years
Population: All patients receiving treatment were evaluated for DLT.
Measure: Number; unit: participants with DLTs
Groups:
- Phase I: Dose Level 1 - Docetaxel 75 mg/m^2: Subjects receive gefitinib 250 mg orally daily, trastuzumab 6 mg/kg intravenously every 3 weeks (after an initial dose of 8 mg/kg with cycle 1), and docetaxel 75 mg/m^2 intravenously every 3 weeks.
- Phase I: Dose Level 2 - Docetaxel 60 mg/m^2: Subjects receive gefitinib 250 mg orally daily, trastuzumab 6 mg/kg intravenously every 3 weeks (after an initial dose of 8 mg/kg with cycle 1), and docetaxel 60 mg/m^2 intravenously every 3 weeks.
Arm/Group | Phase I: Dose Level 1 - Docetaxel 75 mg/m^2 | Phase I: Dose Level 2 - Docetaxel 60 mg/m^2
Number analyzed (Participants) | 2 | 7
participants with DLTs | 2 | 0

2. Primary Outcome: Recommended Phase II Dose
Description: The maximum tolerated dose (MTD): subjects received gefitinib 250 mg orally daily, trastuzumab 6 mg/kg intravenously every 3 weeks (after an initial dose of 8 mg/kg with cycle 1), and docetaxel 75 mg/m^2 intravenously every 3 weeks. This was to serve as the phase II dose if no dose-limiting toxicities (DLTs) occurred in the first three subjects. If one DLT occurred in the first three subjects, another three subjects where to be enrolled at this dose, whereas if two DLTs occurred in the first three subjects, the docetaxel dose was to be decreased to 60 mg/m^2. The study would then be continued only if no more than one patient had a DLT at this dose. Once the dose of docetaxel was established, all further subjects were to be treated at the phase II MTD dose.
Time Frame: 4 weeks from start of treatment, up to 2 years
Population: All patients observed for 21 days while receiving a full course of therapy or who experienced a DLT. Patients withdrawing before completion of the first course, for reasons other than DLT, were replaced.
Measure: Number; unit: mg/m^2
Groups:
- Phase I: All patients enrolled on the Phase I (dose-finding) portion of the study.
Arm/Group | Phase I
Number analyzed (Participants) | 9
mg/m^2 | 60

3. Secondary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or the appearance of new lesions.
Time Frame: Until disease progression, up to 5 years.
Population: All patients treated at the phase II docetaxel dose (7 in the phase I portion, 22 in the phase II portion).
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Dose Level 2 - Docetaxel 60 mg/m^2: Subjects receive gefitinib 250 mg orally daily or 250 mg daily on days 2 through 14 depending on study findings, trastuzumab 6 mg/kg intravenously every 3 weeks (after an initial dose of 8 mg/kg with cycle 1), and docetaxel 60 mg/m2 intravenously every 3 weeks.
Arm/Group | Dose Level 2 - Docetaxel 60 mg/m^2
Number analyzed (Participants) | 29
Months | 12.7 [7.6 to 21.8]

4. Secondary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response Rate defined as percentage of patients achieving a Best Response of either CR or PR.
Time Frame: After 3 cycles of treatment, up to 2 years.
Population: All patients treated at the phase II docetaxel dose (7 in the phase I portion, 22 in the phase II portion). Patients who complete 3 cycles of treatment or who terminate treatment for reasons of toxicity, or who progress prior to the completion of 3 cycles of therapy on the Phase II portion of the study.
Measure: Number; unit: percentage of participants
Groups:
- Dose Level 2 - Docetaxel 60 mg/m^2: Subjects receive gefitinib 250 mg orally daily or 250 mg daily on days 2 through 14 depending on study findings, trastuzumab 6 mg/kg intravenously every 3 weeks (after an initial dose of 8 mg/kg with cycle 1), and docetaxel 60 mg/m^2 intravenously every 3 weeks.
Arm/Group | Dose Level 2 - Docetaxel 60 mg/m^2
Number analyzed (Participants) | 29
percentage of participants | 64

5. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: Until death from any cause, up to 5 years.
Population: All patients treated at the phase II docetaxel dose (7 in the phase I portion, 22 in the phase II portion).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Level 2 - Docetaxel 60 mg/m^2
Number analyzed (Participants) | 29
Months | 43.2 [30.8 to 65.3]

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 5 years and 3 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Groups:
- Dose Level 1 - Docetaxel 75 mg/m^2: Subjects receive gefitinib 250 mg orally daily, trastuzumab 6 mg/kg intravenously every 3 weeks (after an initial dose of 8 mg/kg with cycle 1), and docetaxel 75 mg/m^2 intravenously every 3 weeks.
Arm/Group | Dose Level 1 - Docetaxel 75 mg/m^2 | Dose Level 2 - Docetaxel 60 mg/m^2
Serious Adverse Events (participants affected / at risk) | 2/2 | 7/29
Other Adverse Events (participants affected / at risk) | 2/2 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - Docetaxel 75 mg/m^2 (N=2) | Dose Level 2 - Docetaxel 60 mg/m^2 (N=29)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Haemorrhage NOS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Infection NOS (Infections and infestations) | 0 (0) | 2 (2)
Leukopenia (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - Docetaxel 75 mg/m^2 (N=2) | Dose Level 2 - Docetaxel 60 mg/m^2 (N=29)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (9) | 25 (196)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 9 (18)
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 2 (3)
Left ventricular failure (Cardiac disorders) | 1 (1) | 5 (8)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 3 (3)
Palpitations (Cardiac disorders) | 0 (0) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 8 (24)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (3)
Ear pain (Ear and labyrinth disorders) | 1 (2) | 3 (4)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 1 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 0 (0) | 2 (2)
Eye disorder (Eye disorders) | 0 (0) | 4 (7)
Vision blurred (Eye disorders) | 1 (1) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 8 (18)
Constipation (Gastrointestinal disorders) | 1 (1) | 6 (16)
Diarrhea (Gastrointestinal disorders) | 2 (5) | 26 (129)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (9)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (4)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (2) | 9 (44)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (4) | 15 (32)
Nausea (Gastrointestinal disorders) | 2 (5) | 18 (44)
(Gastrointestinal disorders) | 0 (0) | 2 (8)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 0 (0) | 2 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 11 (17)
Chest pain (General disorders) | 1 (1) | 3 (10)
Chills (General disorders) | 2 (3) | 8 (12)
Edema (General disorders) | 0 (0) | 2 (3)
Fatigue (General disorders) | 2 (3) | 28 (158)
Fever (General disorders) | 0 (0) | 11 (17)
General symptom (General disorders) | 0 (0) | 3 (5)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Oedema NOS (General disorders) | 2 (5) | 6 (9)
Pain (General disorders) | 2 (5) | 16 (60)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 1 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Immune system disorder (Immune system disorders) | 0 (0) | 3 (4)
Infection (Infections and infestations) | 1 (2) | 5 (7)
Infection NOS (Infections and infestations) | 1 (2) | 9 (15)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 1 (1)
Infection without neutropenia (Infections and infestations) | 0 (0) | 3 (3)
Infection, Viral (COH) (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (3)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Intraoperative gastrointestinal injury - Teeth (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 6 (45)
Alanine aminotransferase increased (Investigations) | 1 (2) | 25 (97)
Alkaline phosphatase increased (Investigations) | 1 (1) | 14 (30)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (5) | 25 (150)
Bilirubin increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 4 (4)
Hyperbilirubinemia (Investigations) | 0 (0) | 1 (1)
Hypercholesterolemia (Investigations) | 1 (3) | 1 (1)
INR increased (Investigations) | 2 (4) | 14 (92)
Laboratory test abnormal (Investigations) | 0 (0) | 9 (26)
Leukocyte count decreased (Investigations) | 0 (0) | 12 (65)
Leukopenia (Investigations) | 2 (6) | 16 (103)
Lymphocyte count decreased (Investigations) | 0 (0) | 13 (93)
Lymphopenia (Investigations) | 2 (5) | 12 (107)
Neutrophil count decreased (Investigations) | 2 (4) | 24 (142)
Platelet count decreased (Investigations) | 1 (1) | 5 (5)
Weight gain (Investigations) | 1 (2) | 7 (26)
Weight loss (Investigations) | 1 (3) | 9 (20)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 8 (15)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1) | 5 (6)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 11 (42)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 5 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 13 (53)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 4 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4) | 13 (55)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (5) | 11 (30)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 10 (29)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 9 (22)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 14 (54)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 8 (25)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 6 (8)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 3 (8)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 7 (25)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 6 (15)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 10 (23)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (19)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 5 (10)
Headache (Nervous system disorders) | 1 (2) | 10 (22)
Neuralgia (Nervous system disorders) | 0 (0) | 5 (7)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 6 (7)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 9 (26)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Taste alteration (Nervous system disorders) | 0 (0) | 8 (11)
Anxiety (Psychiatric disorders) | 0 (0) | 10 (13)
Depression (Psychiatric disorders) | 0 (0) | 7 (9)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 1 (1) | 5 (6)
Protein urine positive (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 3 (3)
Reproductive tract disorder (Reproductive system and breast disorders) | 0 (0) | 1 (3)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 12 (36)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 12 (27)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 9 (21)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (24)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 11 (16)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (15)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 9 (9)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (5) | 24 (77)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 12 (30)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (2) | 4 (9)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 2 (3)
Hypertension (Vascular disorders) | 1 (5) | 3 (4)
Hypotension (Vascular disorders) | 1 (1) | 7 (8)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes